CLINICAL TRIAL: NCT02475772
Title: A Phase I, Single-arm, Open-label, Three Step Dose Escalation Study With Intraperitoneal Pressurized Cisplatin and Doxorubicin in Recurrent Ovarian Cancer and Peritoneal Carcinomatosis
Brief Title: A Study With Intraperitoneal Cisplatin and Doxorubicin in Recurrent Ovarian Cancer and Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clemens Tempfer (Other)
Responsible Party: Sponsor-Investigator, Clemens Tempfer, Chairman, Clinic Director, Ruhr University of Bochum
Organization: Ruhr University of Bochum (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIPAC-OV2; 2014-001034-28 (EudraCT Number)
Record Dates: First submitted 2014-03-27; First posted 2015-06-19 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; recurrent; chemotherapy; intraperitoneal; cisplatin; doxorubicin
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Cisplatin; Doxorubicin; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin and doxorubicin (Experimental): Cisplatin and doxorubicin will be applied under pressure into the abdomen via laparoscopic trocars. The first 5 patients will receive doxorubicin 1.5 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 7.5 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. The next 5 patients will receive doxorubicin 2.25 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 11.25 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. The next 5 patients will receive doxorubicin 3 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 15 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. This schedule represents a three-step, 50% dose-escalation. Dose density will not be changed.
  Interventions: Drug: Cisplatin and doxorubicin; Procedure: Cisplatin and doxorubicin

INTERVENTIONS:
Drug: Cisplatin and doxorubicin — The first 5 patients will receive doxorubicin 1.5 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 7.5 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. The next 5 patients will receive doxorubicin 2.25 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 11.25 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. The next 5 patients will receive doxorubicin 3 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 15 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. This schedule represents a three-step, 50% dose-escalation. Dose density will not be changed.
  Other Names: Cisplatin TEVA, Doxorubicin 50 HEXAL®
Procedure: Cisplatin and doxorubicin — intraperitoneal chemotherapy with cisplatin and doxorubicin in a dose-escalation scheme
  Other Names: Intraperitoneal chemotherapy

SUMMARY:
Fifteen women with recurrent ovarian cancer will be treated by an intraperitoneal chemotherapy with cisplatin and doxorubicin in three escalating dosage schedules. The aim of the study is to evaluate the safety and tolerability of doxorubicin and cisplatin every 4 weeks for three courses using a three-group, dose-escalation protocol with fixed dose-density. The time Frame for the assessment of the Primary outcome is therefore 12 weeks. Predefined toxicity criteria will be applied using CTCAE version 4.0 criteria. The study hypothesis is that local and systemic toxicity will increase with increasing dosage of cisplatin and doxorubicin during three repeated PIPAC courses with no CTCAE grade 4 and 5 events in any treatment group.

DETAILED DESCRIPTION:
This is a prospective phase I, single-arm (nonrandomized), open-label, three step dose-escalation study with cisplatin and doxorubicin applied as PIPAC in 15 patients with recurrent ovarian cancer and peritoneal cancer.

The first 5 patients will receive doxorubicin 1.5 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 7.5 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. The next 5 patients will receive doxorubicin 2.25 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 11.25 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. The next 5 patients will receive doxorubicin 3 mg/m2 body surface in 50 ml NaCl 0,9% and cisplatin 15 mg/m2 in 50 ml NaCl 0,9% q 4 weeks for three courses. This schedule represents a three-step, 50% dose-escalation. Dose density will not be changed.

The aim of this study is to evaluate the safety and tolerability of doxorubicin and cisplatin every 4-6 weeks for three courses using a three-group, dose-escalation protocol with fixed dose-density. The time Frame for the assessment of the Primary outcome is therefore 12 weeks. Predefined toxicity criteria will be applied using CTCAE version 4.0 criteria, documented after the first, second, and third course of treatment. Clinical examinations will include abdominal computed tomography (CT) scans after the first, second, and third course of treatment, cardiac echocardiography before the first, second, and third course of treatment, and a clinical neurological assessment before the first, second, and third course of treatment. Pharmacological studies will include hematologic, liver, and renal function tests as well as cisplatin and doxorubicin plasma levels with blood samples drawn before, during, and up to 12 h after the start of each PIPAC course.

ELIGIBILITY:
Inclusion Criteria:

1. clinical and/or radiological evidence of PC,
2. age between 18 and 85 years with a diagnosis of recurrent ovarian cancer with disease progression after at least one line of previous intravenous chemotherapy with a platinum compound,
3. blood and electrolyte counts, liver, and renal function parameters within 10% of the normal range established in the respective laboratory of the study institution,
4. provision of written informed consent, and
5. postmenopausal status.

Exclusion Criteria:

1. extraabdominal metastatic disease, with the exception of isolated pleural carcinomatosis/effusion,
2. chemotherapy or surgery within the last four weeks prior to the first PIPAC application,
3. previous treatment with maximum cumulative doses of doxorubicin, daunorubicin, epirubicin, idarubicin, and/or other anthracyclines and anthracenediones,
4. a history of allergic reaction to cisplatin or other platinum containing compounds or doxorubicin,
5. severe renal impairment, myelosuppression, severe hepatic impairment, severe myocardial insufficiency, recent myocardial infarction or severe cardiac arrhythmia,
6. immunocompromised status such as immunosuppressive therapy or a known disease of the immune system,
7. previous enrolment in the present study, and
8. previous intraabdominal chemotherapy or intraabdominal antibody therapy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Adverse events according to CTCAE criteria | 12 weeks

SECONDARY OUTCOMES:
Clinical benefit according to RECIST criteria | 12 weeks

OTHER OUTCOMES:
Plasma concentrations of cisplatin and doxorubicin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clemen^s B Tempfer, MD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Ruhr University Bochum, Germany, Marienhospital Herne, Herne, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Tempfer CB, Celik I, Solass W, Buerkle B, Pabst UG, Zieren J, Strumberg D, Reymond MA. Activity of Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) with cisplatin and doxorubicin in women with recurrent, platinum-resistant ovarian cancer: preliminary clinical experience. Gynecol Oncol. 2014 Feb;132(2):307-11. doi: 10.1016/j.ygyno.2013.11.022. Epub 2013 Nov 23. PMID 24275155
- [Result] Tempfer CB, Giger-Pabst U, Seebacher V, Petersen M, Dogan A, Rezniczek GA. A phase I, single-arm, open-label, dose escalation study of intraperitoneal cisplatin and doxorubicin in patients with recurrent ovarian cancer and peritoneal carcinomatosis. Gynecol Oncol. 2018 Jul;150(1):23-30. doi: 10.1016/j.ygyno.2018.05.001. Epub 2018 May 6. PMID 29743140